CLINICAL TRIAL: NCT01790724
Title: Social Cognitive and Neuropsychological Influences on Physical Activity Behavior in Type II Diabetes
Brief Title: Regulating Efficacy and Wellness in Diabetes
Acronym: REWinD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Edward McAuley, Principal Investigator, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13146; 1F31AG042232-01A1 (NIH)
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Type 2; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walking exercise (Experimental): Participants will be instructed in safe walking exercise. They will participate in an eight week, tapered, on-site program. Participants will also attend group workshops where they will learn self-regulatory skills such as goal-setting, self-monitoring, barrier trouble-shooting, rewarding, and relapse prevention and recovery.
  Interventions: Behavioral: Walking exercise
- Metabolic health education (Active Comparator): Participants will complete an eight-week online metabolic health education course. Topics will include glucose control, insulin, weight management, nutrition, physical activity, eye/kidney/foot health, stress reduction, and doctor-patient communication.
  Interventions: Behavioral: Walking exercise

INTERVENTIONS:
Behavioral: Walking exercise

SUMMARY:
The propose of the study is to test the hypothesis that an eight week program consisting of walking exercise and social cognitive theory based group workshops will increase physical activity adherence six months later in older adults with type 2 diabetes or metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* adults between the ages of 50-75 years
* individuals diagnosed with type 2 diabetes or metabolic syndrome (presence of 3 of the 5 criteria)
* physician consent to participate.

Exclusion Criteria:

* below age 50 or above age 75 at the beginning of the intervention
* exercising regularly more than twice per week for the last six months
* diagnosis of type 1 diabetes mellitus
* failing the Telephone Interview of Cognitive Status
* inability to communicate in English

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Month 6
  Change from baseline to month six in physical activity. Participants will wear an accelerometer to measure physical activity.

SECONDARY OUTCOMES:
Self-efficacy | Month 6
  We will assess changes in self-efficacy by written questionnaires.
Executive function | Month 6
  Participants will complete a neuropsychological battery of tasks assessing memory, attention and decision-making at baseline and month six.
Self-regulatory strategy use | Month 6
  We will assess changes in self-regulatory strategy use by written questionnaires.
Physical function | Month 6
  We will conduct functional fitness testing including tests of balance, strength, mobility and flexibility at baseline and six months.
Psychosocial outcomes | Month 6
  We will assess changes in psychosocial function ( e.g. self-esteem; social support; anxiety) by written questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Edward McAuley, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

REFERENCES:
- [Derived] Olson EA, Mullen SP, Raine LB, Kramer AF, Hillman CH, McAuley E. Integrated Social- and Neurocognitive Model of Physical Activity Behavior in Older Adults with Metabolic Disease. Ann Behav Med. 2017 Apr;51(2):272-281. doi: 10.1007/s12160-016-9850-4. PMID 27844326
- See also: Exercise Psychology Lab at University of Illinois at Urbana-Champaign — http://www.epl.illinois.edu